CLINICAL TRIAL: NCT05227313
Title: Evaluation Dietary Supplement" Eefooton" on the Quality of Life in Chronic Kidney Disease
Brief Title: Double-Blind, Placebo-Controlled Trial of Eefooton in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Collaborators: Morris Enterprise Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB No.10-FS-088
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases; Renal Insufficiency, Chronic; Urologic Diseases
Keywords: eGFR; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Urologic Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eefooton oral solution (Experimental): 20ml, 3 times per day (daily dose: 60 ml)
  Interventions: Dietary Supplement: Eefooton oral solution; Dietary Supplement: Placebo oral solution
- Placebo oral solution (Placebo Comparator): oral solution matched placebo
  Interventions: Dietary Supplement: Eefooton oral solution; Dietary Supplement: Placebo oral solution

INTERVENTIONS:
Dietary Supplement: Eefooton oral solution — Eefooton is extracted from Rhodiola, Huang Qi, American Ginseng, Dang Ginseng, and Ligustrum lucidum by biotechnology. It has immunomodulatory effects, anti-oxidation and anti-inflammatory effects, and regulates calcium metabolism.
Dietary Supplement: Placebo oral solution — oral solution matched placebo

SUMMARY:
This phase II study, 24-week, double-blind, study evaluated Eefooton's safety and efficacy for patients with CKD stage 3 to 4 Not on dialysis.

DETAILED DESCRIPTION:
The purpose of this clinical observation and research is to evaluate the eGFR changes in the renal function of patients with chronic kidney disease combination the Eefooton oral solution and commonly used chemical drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic kidney disease who have signed the subject's consent and the glomerular filtration rate (eGFR) is less than 59ml/min/1.73m2
2. Both male and female patients aged 20-85 years old are acceptable
3. You must be able to come back at a specific time each month during the 6-month trial

Exclusion Criteria:

1. Drug abuse.
2. Heart failure (stage 3-4)
3. Mental illness (psychotic disorder, epilepsy, depression, panic disorder)
4. Patients who have undergone dialysis or are expected to have a kidney transplant in the last three months
5. The blood pressure still exceeds 150/90mmHg after using more than three antihypertensive drugs
6. Pregnancy or planning to become pregnant or breastfeeding
7. Malignant disease
8. Acute illness (hepatitis, jaundice, acute myocardial infarction) in the last 3 months
9. The patient is engaged in another research study.
10. 3 months before entering the study or having used NSAIDs, anti-rejection drugs or performing imaging agent examinations during the study
11. You have participated in other research study in the previous month
12. You have drug dependence and drinking habits

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Short-Form 36 Questionnaire | 2month
  The SF-36 questionnaire consists of eight health concepts, each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. (1) physical functioning, (2) role limitations due to physical health, (3) bodily pain, (4) general health perceptions, (5) vitality (energy/fatigue), (6) social functioning, (7) role limitations due to emotional health, (8) general mental health

SECONDARY OUTCOMES:
eGFR value | one month
  The eGFR value is an important marker for kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Cheng Lu, Ph.D, Study Chair — Taichung Tzu Chi Hospital; Chen-Shiung Wu, Ph.D, Study Director — Taichung Tzu Chi Hospital; Ching-Hsiu Peng, MD, Principal Investigator — Taichung Tzu Chi Hospital; Ko-Lin Kuo, MD, Principal Investigator — Taichung Tzu Chi Hospital; Yi-Chun Wang, MD, Principal Investigator — Taichung Tzu Chi Hospital; Ding-Jun Lin Lin, MD, Principal Investigator — Taichung Tzu Chi Hospital; Szu-Chun Hung, MD, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Department of Nephrology, Taipei Tzu Chi Hospital, Taipei, Taiwan, Taipei County, Taiwan